CLINICAL TRIAL: NCT06988826
Title: Comparison of Antibiotics With and Without Granulocyte Colony-Stimulating Factor in Children With Chemotherapy Induced Febrile Neutropenia
Brief Title: Comparison of G-CSF & Antibiotics Versus Antibiotics Alone in Resolution of Febrile Neutropenia
Acronym: AGF-FN
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: King Edward Medical University (Other)
Collaborators: University of Child Health Sciences and Children's Hospital, Lahore (Other)
Responsible Party: Principal Investigator, Sidrah Lodhi, Assistant Professor of Endocrinology, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 656/CH-UCHS/15/5/2023
Record Dates: First submitted 2025-05-14; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Febrile Neutropenia; Febrile Neutropenia, Rule of Clinical Decision, Chemotherapy; Febrile Neutropenia, Drug-Induced; G-CSF; Antibiotic Therapy
Keywords: febrile neutropenia; chemotherapy-induced febrile neutropenia; Antibiotics; G-CSF
MeSH Terms: conditions — Febrile Neutropenia; Chemotherapy-Induced Febrile Neutropenia | interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): G-CSF plus antibiotic therapy
  Interventions: Drug: G-CSF
- Group 2 (Active Comparator): Antibiotic Therapy
  Interventions: Drug: Antibiotics only

INTERVENTIONS:
Drug: G-CSF — G-CSF & Antibiotic therapy in combination
  Arms: Group 1
Drug: Antibiotics only — Antibiotics alone
  Arms: Group 2

SUMMARY:
This study aim to find the best option for children having cancer who develop low immunity state due to chemotherapy

DETAILED DESCRIPTION:
Children having a cancer diagnosis and treated with chemotherapy often develop neutropenia. This creates an immunocompromised state which can result in infections manifested by fever. This study compares two treatment options to find out the best treatment for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-16 years
* any Gender
* Febrile neutropenia
* diagnosed case of solid or hematological malignancy
* taking chemotherapy

Exclusion Criteria:

* Non-neutropenic fever
* already received G-CSF or antibiotics before presenting to hospital
* any other cause of neutropenia

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Resolution of FN | 2 weeks
  Duration of resolution of febrile neutropenia (in days)

SECONDARY OUTCOMES:
Afebrile | 2 weeks
  Duration of resolution of fever (in days)
Length of hospital stay | 2 weeks
  Length of hospital stay (in days)

IPD SHARING:
Plan to Share IPD: Yes
Data dictionary will be made available on request
Supporting Information: Study Protocol